CLINICAL TRIAL: NCT02395250
Title: Autologous T Cells Redirected to GPC3 for Treating Patients With Advanced HCC
Brief Title: Anti-GPC3 CAR T for Treating Patients With Advanced HCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-20150313
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2018-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anti-GPC3 CAR T (Experimental)
  Interventions: Biological: anti-GPC3 CAR T

INTERVENTIONS:
Biological: anti-GPC3 CAR T
  Other Names: CAR T cells redirected to Glypican-3 in cancer cells

SUMMARY:
The purpose of this study is to determine whether autologous T cells bearing chimeric antigen receptor that can specifically recognize glypican-3 (GPC3) is safe and effective for patients with relapsed or refractory hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion criteria:

1. Age of 18-70 years;
2. Pathologically confirmed advanced hepatocellular carcinoma (HCC);
3. ≥1 measurable target lesion per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1);
4. Tumor tissue positive for GPC3 expression per immunohistochemical staining (IHC) assay;
5. Estimated survival > 12 weeks;
6. Child-Pugh grade A;
7. ECOG performance score of 0-1;
8. HBV-DNA < 200 IU/mL if positive for HBsAg or HBcAb. Patients positive for HBsAg shall receive anti-viral treatment per "The guideline of prevention and treatment for chronic hepatitis B: a 2015 update";
9. Have adequate venous access for apheresis or venous blood collection;
10. White blood cells ≥ 2.5 x 109/L, platelet ≥ 60×109/L, haemoglobin ≥ 9.0 g/dL, lymphocyte ≥ 0.4×109/L
11. Serum albumin ≥ 30 g/dL, serum lipase and amylase≤1.5 upper limit of normal (ULN), serum creatinine ≤ 1.5 ULN and endogenous creatinine clearance ≥ 40mL/min, ALT and AST ≤ 5 ULN, Serum total bilirubin ≤ 2.5 ULN, Prothrombin Time is less than 4s longer than normal;
12. Negative serum pregnancy test within 14 days before CAR T infusion, and with willingness to use reliable contraceptive methods to avoid pregnancy until 12 months after CAR T infusions for females of childbearing age; Having undergone sterilization procedure or with willingness to use reliable contraceptive methods to avoid pregnancy for males with female partner of childbearing age during the study;
13. Able to understand and sign the informed consent form

Exclusion criteria:

If the patient meets any of the exclusion criteria, the patient must be excluded from the study.

1. Pregnant or lactating female patients;
2. Positive serum tests for HCV, HIV, or syphilis;
3. Presence of HBV/HCV coinfection;
4. Presence of any uncontrollable active infection, such as, but not limited to, active tuberculosis
5. History of systemic administration of steroids (not including inhaled steroids), or other immunosuppressant drugs within 2 weeks before apheresis;
6. History of allergy to immunotherapy and related drugs, or β-lactam antibiotics, or history of other severe allergy;
7. History or current presence of hepatic encephalopathy;
8. Presence of ascites with clinical significance that is defined as positive focused physical examination for ascites, or ascites that requires treatment intervention (not including any ascites shown on image examinations without the need for clinical intervention);
9. ≥ 50% of normal liver occupied with HCC tumor tissue, or presence of tumor thrombus in the portal vein, or mesenteric vein, or inferior vena based on image analysis;
10. Presence of HCC metastatic lesion in the central nervous system, or presence of other diseases of central nervous system with clinical significance;
11. Presence of heart disease that requires treatment intervention, or poorly controlled hypertension (systolic pressure > 160 mmHg, or diastolic pressure > 100 mmHg);
12. Presence of active auto-immune disease that requires immunosuppressant treatment;
13. History of organ transplantation or currently on the waiting list for organ transplantation, including, but not limited to, liver transplantation;
14. Anti-HCC therapies including, but not limited to, surgical resection, interventional therapy, radiation therapy, chemotherapy, and immunotherapy, within 2 weeks before apheresis;
15. History of receiving anti-PD-1 or anti-PD-L1 monoclonal antibodies, or other immunotherapy;
16. History of other malignancies in the past 5 years, or presence of other active malignancies (not including cervical cancer in situ and basal cell carcinomas);
17. Presence of other serious diseases or conditions, including uncontrolled diabetes (HbA1c > 7% with treatment); severe cardiac dysfunction with LVEF < 45%; myocardial infarction, unstable angina, or unstable arrhythmia in the past 6 months pulmonary embolism; chronic obstructive pulmonary disease; interstitial lung disease; forced expiratory volume in 1 second (FEV1) < 60%, gastric ulcer; history of gastrointestinal bleeding, or confirmed tendency for gastrointestinal bleeding;
18. Determined by the investigator to be lack of compliance for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Adverse events attributed to the administration of the anti-GPC3 CAR T cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhai, MD, Study Director — Renji
Locations (1):
- Shanghai Cancer Institute, Xuhui, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Shi D, Chi J, Cui D, Tang X, Lin Y, Wang S, Li Z, Jin H, Zhai B. Combined local therapy and CAR-GPC3 T-cell therapy in advanced hepatocellular carcinoma: a proof-of-concept treatment strategy. Cancer Commun (Lond). 2023 Sep;43(9):1064-1068. doi: 10.1002/cac2.12472. Epub 2023 Jul 21. No abstract available. PMID 37478283